CLINICAL TRIAL: NCT06278129
Title: Evaluation of the Diagnostic and Prognostic Efficacy of Magnetic Resonance Imaging in Patients With Acute Sensorineural Hearing Loss and Ménière's Disease
Brief Title: Evaluation of the Diagnostic and Prognostic Efficacy of MRI in Acute Sensorineural Hearing Loss and Ménière's Disease
Acronym: MRI_SSHL/MD
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 4146
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Sudden Sensorineural Hearing Loss; Meniere Disease; Ménière's Vertigo; Meniere's Disease Aggravated; Inner Ear Disease
MeSH Terms: conditions — Hearing Loss, Sudden; Meniere Disease; Labyrinth Diseases | interventions — Vestibular Evoked Myogenic Potentials; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Vestibular myogenic potentials — observational study
  Other Names: Magnetic resonance imaging

SUMMARY:
Evaluation of the diagnostic and prognostic efficacy of nuclear magnetic resonance imaging in patients with acute sensorineural hearing loss or in patients suffering from probable or definite MD. The neuroradiological and audiological evaluation are held on in the same day in order to better clarify the radiological and clinical correlates.

DETAILED DESCRIPTION:
Aims of the study:

1. Evaluate the diagnostic accuracy of MRI with the collection of more specific sequences for the inner ear (3D-FLAIR) in identifying intralabyrinthine anomalies in patients with Ménière's disease or acute/subacute sudden hearing loss and not only the retrochlear pathology/neurological causes .
2. Characterize the vascular and inflammatory MRI patterns
3. Define the prognostic role of MRI with pre- and post-contrast 3D-FLAIR sequence, eliminating confounding factors such as MRI execution time, the methodology used, the effect of previous therapy and the criteria for defining improvement.
4. Correlate 4-hour 3D-FLAIR MRI imaging data with clinical and hematological data

ELIGIBILITY:
Inclusion Criteria:

age > 18 years

* onset of symptoms less than 10 days
* no previous episodes of sudden ipsilateral hearing loss
* no systemic or oral corticosteroid intake in the previous month
* Informed consent

Exclusion Criteria:

* Current or previous otopathy and/or labyrinth diseases of known cause
* Known nervous system disorders
* Patients with renal insufficiency (creatinine level > 1.5 mg/dL)
* Patients with pacemakers, other metal implants, claustrophobics and known psychiatric disorders
* Pregnant patients Materials and methods Diagnostic evaluation at enrollment (T0)
* Audiological or ENT examination
* Liminal tonal audiometric exam, vocal, impedance measurement, otoacoustic emissions, video-impulse test, oVEMPS, cVEMPS, stabilometry
* Hematological tests: complete blood count, ESR, PCR, creatininemia, CMV IgM, EBV IgM, ANA, glycemia, study of predisposing genetic factors

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients suffering from acute sudden hearing loss and Meniere's disease according to the criteria of the American Academy of Otolaryngology.
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2018-06-19 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of inner ear structures in MRI images | 1 day
  MRI - ocular and cervical VEMPS - audiological and otoneurological evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Audiology and Neuroradiology - Milan (Italy), Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Conte G, Di Berardino F, Sina C, Zanetti D, Scola E, Gavagna C, Gaini L, Palumbo G, Capaccio P, Triulzi F. MR Imaging in Sudden Sensorineural Hearing Loss. Time to Talk. AJNR Am J Neuroradiol. 2017 Aug;38(8):1475-1479. doi: 10.3174/ajnr.A5230. Epub 2017 May 25. PMID 28546251
- [Background] Conte G, Caschera L, Calloni S, Barozzi S, Di Berardino F, Zanetti D, Scuffi C, Scola E, Sina C, Triulzi F. MR Imaging in Meniere Disease: Is the Contact between the Vestibular Endolymphatic Space and the Oval Window a Reliable Biomarker? AJNR Am J Neuroradiol. 2018 Nov;39(11):2114-2119. doi: 10.3174/ajnr.A5841. Epub 2018 Oct 18. PMID 30337432
- [Background] Conte G, Di Berardino F, Zanetti D, Avignone S, Sina C, Iofrida E, Triulzi F. The 'full-blown' MRI of sudden hearing loss: 3D FLAIR in a patient with bilateral metastases in the internal auditory canals. Neuroradiol J. 2018 Feb;31(1):39-41. doi: 10.1177/1971400917736927. Epub 2017 Oct 19. PMID 29046124
- [Background] Berardino FD, Conte G, Turati F, Ferraroni M, Zanetti D. Cochlear implantation in Meniere's disease: a systematic review of literature and pooled analysis. Int J Audiol. 2020 Jun;59(6):406-415. doi: 10.1080/14992027.2020.1720922. Epub 2020 Feb 6. PMID 32027195
- [Background] Conte G, Lo Russo F, Caschera L, Zanetti D, Castorina P, Sina C, Triulzi F, Di Berardino F. Audiovestibular Phenotypes and Advanced Magnetic Resonance Imaging Features of Cochlin Gene Mutation Carriers. Audiol Neurootol. 2019;24(4):166-173. doi: 10.1159/000501292. Epub 2019 Aug 7. PMID 31390618
- [Result] Conte G, Di Berardino F, Zanetti D, Iofrida EF, Scola E, Sbaraini S, Filipponi E, Cinnante C, Gaini LM, Ambrosetti U, Triulzi F, Pignataro L, Capaccio P. Early Magnetic Resonance Imaging for Patients With Idiopathic Sudden Sensorineural Hearing Loss in an Emergency Setting. Otol Neurotol. 2019 Oct;40(9):1139-1147. doi: 10.1097/MAO.0000000000002389. PMID 31498290
- [Result] Conte G, Di Berardino F, Mastrapasqua RF, Casale S, Scola E, Capaccio P, Triulzi F, Pignataro L, Zanetti D. Prognostic Value of Early Magnetic Resonance Imaging Patterns in Sudden Hearing Loss. Audiol Neurootol. 2022;27(1):64-74. doi: 10.1159/000515153. Epub 2021 Apr 23. PMID 33895732